CLINICAL TRIAL: NCT00002236
Title: An Open-Label, Parallel Group, Pilot Study of Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of BID and TID Regimens of Delavirdine Mesylate, Zidovudine, and Indinavir Sulfate in HIV-1 Infected Individuals
Brief Title: A Study to Find the Best Dosing Schedule for Delavirdine, Zidovudine, and Indinavir in HIV-Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 228G; M/3331/0072
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; Drug Administration Schedule; HIV Protease Inhibitors; CD4 Lymphocyte Count; Indinavir; Delavirdine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Delavirdine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Delavirdine mesylate
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see whether it is better to take delavirdine (DLV) plus indinavir (IDV) plus zidovudine (ZDV) twice a day or three times a day.

DETAILED DESCRIPTION:
Patients are divided into 2 treatment groups; the groups are balanced with respect to viral load. Group A receives ZDV, DLV, and IDV 3 times daily. Group B receives ZDV, DLV, and IDV 2 times daily. Patients are evaluated for changes from baseline in viral load and CD4 cell count.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a viral load (level of HIV in the blood) of at least 20,000 copies/ml.
* Have a CD4 cell count of at least 50 cells/mm3.
* Are at least 14 years old (consent of parent or guardian is required if under 18).

Exclusion Criteria

You will not be eligible for this study if you:

* Have ever taken an anti-HIV drug other than ZDV.
* Have taken ZDV for more than 1 month.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - AIDS Healthcare Foundation, Los Angeles, California
  - UCSF AIDS Research Institute, San Francisco, California
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Univ of Tennessee / Div of Infect Dis / Dept of Med, Memphis, Tennessee
  - Infectious Disease Physicians Inc, Annandale, Virginia